CLINICAL TRIAL: NCT03730194
Title: A SMART Design to Improve Sleep Disturbance in Adolescents With Neurodevelopmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 0775-18-FB; 1K01NR017465-01A1 (NIH)
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Results first posted 2023-04-04 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Sleep Disturbance
Keywords: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Sleep Disturbance; Melatonin; ASD; ADHD
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Parasomnias | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: The investigators utilized a sequential, multiple assignment, randomized trial (SMART) pilot feasibility study design to inform implementation of a future full-scale SMART design that will be used to construct adaptive biobehavioral sleep intervention strategies involving melatonin, a behavioral sleep intervention (The Bedtime Bank), and their combination for the management of sleep disturbance in adolescents with neurodevelopmental (NDDs). Participants completed 1 week of baseline data collection, and than were randomly assigned to either melatonin or The Bedtime Bank. Response (>/= 18 minute average nightly increase in total sleep time [TST]) was measured at Week 4 and Week 8. Participants who responded (>/= 18 minute average nightly increase in TST) at Week 4 remained on the assigned intervention. Participants who were non-responsive at Week 4 were re-randomized to a different sleep intervention or combined interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Melatonin Only (Experimental): In stage 1, participants in this arm will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
  In stage 2, responders to melatonin will take 3 mg of melatonin 30 minutes before bedtime for an additional 4 weeks (repeat stage 1, for a total of 8 weeks).
  Interventions: Dietary Supplement: Melatonin
- The Bedtime Bank Only (Experimental): In stage 1, participants in this arm will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  In stage 2, responders to The Bedtime Bank will utilize The Bedtime Bank, a behavioral sleep intervention for an additional 4 weeks (repeat stage 1, for a total of 8 weeks).
  Interventions: Behavioral: Bedtime Bank
- Melatonin than Bedtime Bank (Experimental): In stage 1, participants in this arm will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
  In stage 2, non-responders to melatonin will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  Interventions: Dietary Supplement: Melatonin; Behavioral: Bedtime Bank
- Melatonin than Melatonin+Bedtime Bank Combo (Experimental): In stage 1, participants in this arm will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
  In stage 2, non-responders to melatonin will take 3 mg of melatonin 30 minutes before bedtime for an additional 4 weeks (repeat stage 1, for a total of 8 weeks) AND utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  Interventions: Dietary Supplement: Melatonin; Behavioral: Bedtime Bank
- Bedtime Bank than Melatonin (Experimental): In stage 1, participants in this arm will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  In stage 2, non-responders to The Bedtime Bank will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
  Interventions: Dietary Supplement: Melatonin; Behavioral: Bedtime Bank
- Bedtime Bank than Bedtime Bank+Melatonin Combo (Experimental): In stage 1, participants in this arm will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  In stage 2, non-responders to The Bedtime Bank will utilize The Bedtime Bank, a behavioral sleep intervention for an additional 4 weeks (repeat stage 1, for a total of 8 weeks) AND take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
  Interventions: Dietary Supplement: Melatonin; Behavioral: Bedtime Bank

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin (liquid, immediate release, 3 mg) 30 minutes before bedtime
  Arms: Bedtime Bank than Bedtime Bank+Melatonin Combo; Bedtime Bank than Melatonin; Melatonin Only; Melatonin than Bedtime Bank; Melatonin than Melatonin+Bedtime Bank Combo
Behavioral: Bedtime Bank — The Bedtime Bank a novel behavioral sleep intervention, which is based upon contingency contracting and relies on a credit or debt-based system to hold adolescents accountable for maintaining a consistent bedtime and improve total sleep time.
  Arms: Bedtime Bank than Bedtime Bank+Melatonin Combo; Bedtime Bank than Melatonin; Melatonin than Bedtime Bank; Melatonin than Melatonin+Bedtime Bank Combo; The Bedtime Bank Only

SUMMARY:
The objective of this K01 study was to pilot a sequential, multiple assignment, randomized trial (SMART) design to compare the impact of a sequence of sleep interventions, based on participant treatment response, to optimize sleep health in adolescents 10-18 years of age with neurodevelopmental disorders (NDDs).

DETAILED DESCRIPTION:
The investigators conducted a sequential, multiple assignment, randomized trial (SMART) pilot feasibility study to inform implementation of a future full-scale SMART design that will be used to construct adaptive biobehavioral sleep intervention strategies involving melatonin, a behavioral sleep intervention (The Bedtime Bank), and their combination for the management of sleep disturbance in adolescents with neurodevelopmental (NDDs). Participants completed 1 week of baseline data collection, and than were randomly assigned to either melatonin or The Bedtime Bank. Response (>/= 18 minute average nightly increase in total sleep time [TST]) was measured at Week 4 and Week 8. Participants who responded (>/= 18 minute average nightly increase in TST) at Week 4 remained on the assigned intervention. Participants who were non-responsive at Week 4 were re-randomized to a different sleep intervention or combined interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-18 years and consistently living with parental (or legal guardian) supervision.
* Diagnostic report of confirmed NDD diagnosis (ASD or ADHD).
* Documentation of adolescent being classified as non-intellectually impaired (e.g. IQ>70).
* Parent report of adolescent spending less than or equal to 8 hours in bed per night on 3 or more nights per week in the past month or a composite score greater than 41 on the Children's Sleep Habits Questionnaire.
* Medication-free or on a stable dose of medications (no changes within 30 days prior to enrollment) with parental agreement to avoid changes in current medication (unless provider directed) during study participation.

Exclusion Criteria:

* Unwillingness to stop melatonin 2 months prior to enrollment in the study.
* Parent report of adolescent with a known sleep disorder (e.g. sleep apnea).
* Adolescents who are not able to take oral medication.
* Adolescents who are visually impaired with known inability to detect light.
* Adolescents with an NDD with known genetic etiology (e.g. Angelman syndrome).
* Unwillingness to wear actigraph daily and complete daily sleep diary throughout the 9-week trial.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson E Hanish, PhD, MSN, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Center for Nursing Science, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almirall D, Compton SN, Gunlicks-Stoessel M, Duan N, Murphy SA. Designing a pilot sequential multiple assignment randomized trial for developing an adaptive treatment strategy. Stat Med. 2012 Jul 30;31(17):1887-902. doi: 10.1002/sim.4512. Epub 2012 Mar 22. PMID 22438190
- [Background] Gruber R, Somerville G, Bergmame L, Fontil L, Paquin S. School-based sleep education program improves sleep and academic performance of school-age children. Sleep Med. 2016 May;21:93-100. doi: 10.1016/j.sleep.2016.01.012. Epub 2016 Feb 15. PMID 27448478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: See uploaded study protocol that includes recruitment details.
Groups:
- Bedtime Bank Only: In stage 1, participants in this arm will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  In stage 2, responders to The Bedtime Bank will utilize The Bedtime Bank, a behavioral sleep intervention for an additional 4 weeks (repeat stage 1, for a total of 8 weeks).
- Melatonin Then Bedtime Bank: In stage 1, participants in this arm will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
  In stage 2, non-responders to melatonin will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
- Melatonin Then Melatonin+Bedtime Bank Combo: In stage 1, participants in this arm will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks
  In stage 2, non-responders to melatonin will take 3 mg of melatonin 30 minutes before bedtime for an additional 4 weeks (repeat stage 1, for a total of 8 weeks) AND utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
- Bedtime Bank Then Melatonin: In stage 1, participants in this arm will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  In stage 2, non-responders to The Bedtime Bank will take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
- Bedtime Bank Then Bedtime Bank+Melatonin Combo: In stage 1, participants in this arm will utilize The Bedtime Bank, a behavioral sleep intervention, for 4 weeks.
  In stage 2, non-responders to The Bedtime Bank will utilize The Bedtime Bank, a behavioral sleep intervention for an additional 4 weeks (repeat stage 1, for a total of 8 weeks) AND ill take 3 mg of melatonin 30 minutes before bedtime for 4 weeks.
Period: First Stage Treatment
Arm/Group | Melatonin Only | Bedtime Bank Only | Melatonin Then Bedtime Bank | Melatonin Then Melatonin+Bedtime Bank Combo | Bedtime Bank Then Melatonin | Bedtime Bank Then Bedtime Bank+Melatonin Combo
Started | 20 | 20 | 0 | 0 | 0 | 0
Completed (This study utilizes a SMART Design. 1 participant from the "Melatonin Only" group withdrew from the study. 1 participant from the "Bedtime Bank Only" group withdrew from the study. 3 participants in the "Melatonin Only" group & 3 participants in the "Bedtime Bank Only" group did not complete all study requirements (e.g., minimum actigraph days). These 6 participants remained in the pilot SMART study (did not want to withdraw), and repeated there assigned treatment in the Second Stage.) | 16 | 16 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 3 | 0 | 0 | 0 | 0
Period: Second Stage Treatment
Arm/Group | Melatonin Only | Bedtime Bank Only | Melatonin Then Bedtime Bank | Melatonin Then Melatonin+Bedtime Bank Combo | Bedtime Bank Then Melatonin | Bedtime Bank Then Bedtime Bank+Melatonin Combo
Started | 7 (** 3 participants did not complete all study requirements during the first stage intervention (noted as protocol violation). Melatonin intervention repeated.) | 5 (** 3 participants did not complete all study requirements during the first stage intervention (noted as protocol violation). The Bedtime Bank intervention repeated.) | 6 | 6 | 7 | 7
Completed | 7 | 5 | 6 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This trial is a pilot SMART design. At the first stage randomization participants were randomly assigned to "Melatonin" Only or "Bedtime Bank Only". The "Combination" intervention is not an option until the second stage randomization.
Groups:
- First Stage Melatonin: Stage 1: Participants in this arm will take 3 mg of melatonin 30 minutes before bedtime.
  Melatonin: Melatonin (liquid, immediate release, 3 mg) 30 minutes before bedtime
- First Stage Bedtime Bank: Stage 1: Participants in this arm will utilize the Bedtime Bank, a behavioral sleep intervention.
  Bedtime Bank: The Bedtime Bank a novel behavioral sleep intervention, which is based upon contingency contracting and relies on a credit or debt-based system to hold adolescents accountable for maintaining a consistent bedtime and improve total sleep time.
- Total: Total of all reporting groups
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.45 (2.95) | 13.00 (2.05) | 13.23 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 16 | 17 | 33
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Diagnosis [Count of Participants; unit: Participants]
  Autism (with or without ADHD) | 3 | 6 | 9
  ADHD only | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Actigraphy (Total Sleep Time)
Description: Objective measure of sleep patterns based on the correlation between sleep-wake state and motor activity. A sleep diary was utilized to guide data analysis.
Time Frame: To be worn daily for the entirety of the study (9 weeks total). Data Reported on First Stage Randomization of Melatonin vs. Bedtime Bank (Data Collected at: Baseline, Week 4, and Week 8)
Population: Data Reported on First Stage Randomization of Melatonin vs. Bedtime Bank (Data Collected at: Baseline, Week 4, and Week 8). Data was analyzed based on first stage randomization regardless of whether participants were responders or non-responders.
Measure: Mean (Standard Deviation); unit: Time (hours.minutes of nightly sleep)
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank
Number analyzed (Participants) | 19 | 20
Time (hours.minutes of nightly sleep)
  Baseline | 7.08 (0.50) | 7.03 (1.01)
  Week 4 | 7.16 (0.42) | 7.01 (0.38)
  Week 8 | 7.06 (0.45) | 7.29 (0.48)

2. Primary Outcome: AARP- Abbreviated Acceptability Rating Profile
Description: Parents completed the Abbreviated Acceptability Rating Profile (AARP), which will be used to indicate minimal treatment acceptability. Parent(s) and adolescent completed a semi-structured interview to discuss treatment acceptability.
  Min/Max Values: 8-48 Higher scores=more acceptable/better
Time Frame: Data Reported on First Stage Randomization of Melatonin vs. Bedtime Bank (Data Collected at: Week 4 and Week 8)
Population: Data Reported on First Stage Randomization of Melatonin vs. Bedtime Bank (Data Collected at: Week 4 and Week 8). Data was analyzed based on first stage randomization regardless of whether participants were responders or non-responders.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank
Number analyzed (Participants) | 19 | 18
units on a scale
  Week 4 | 38.84 (7.19) | 34.00 (6.36)
  Week 8 | 38.84 (6.83) | 37.89 (5.49)

3. Secondary Outcome: Urinary Melatonin
Description: The Genway Biotech Melatonin ELISA Kit (San Diego, CA) will allow for the analysis and quantification of endogenous melatonin.
Time Frame: Completed once during the baseline week prior to first stage randomization. Results reported by first stage randomization group.
Population: First morning void urinary 6-sulphatoxymelatonin (Urine 6SM). Urine 6SM concentrations were expressed in ng per mg of creatinine (ng/mg Cr) to control for renal function and dilution of urine.
Measure: Mean (Standard Deviation); unit: ng/mg Cr
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank
Number analyzed (Participants) | 19 | 20
ng/mg Cr | 81.90 (43.67) | 78.58 (31.50)

4. Secondary Outcome: PROMIS Pediatric Item Bank Sleep Related Impairment
Description: An 8-item questionnaire used to measure self-reported alertness, sleepiness, tiredness, and functional impairments associated with sleep problems during waking hours.
  PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S. general population). Higher scores=worse sleep related impairment
Time Frame: Baseline, Week 4, & Week 8-PROMIS Pediatric Item Bank Sleep Related Impairment t-score.
Population: Baseline, Week 4, & Week 8-PROMIS Pediatric Item Bank Sleep Related Impairment t-score. Data was analyzed based on first stage randomization regardless of whether participants were responders or non-responders.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank
Number analyzed (Participants) | 20 | 20
T-score
  Baseline | 58.73 (2.2) | 58.37 (2.3)
  Week 4: number analyzed (Participants) | 19 | 19
  Week 4 | 53.87 (2.74) | 53.56 (2.8)
  Week 8: number analyzed (Participants) | 19 | 19
  Week 8 | 52.76 (2.7) | 51.62 (2.9)

5. Secondary Outcome: PROMIS Pediatric Item Bank Sleep Disturbance
Description: An 8-item questionnaire used to measure self-reported perceptions of sleep quality, depth, and restoration. This includes perceived difficulties getting to sleep and staying asleep, as well as sleep satisfaction.
  PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S. general population). Higher scores=worse sleep disturbance
Time Frame: Baseline, Week 4, & Week 8 PROMIS Pediatric Item Bank Sleep Disturbance t-scores/SE.
Population: Baseline, Week 4, & Week 8 PROMIS Pediatric Item Bank Sleep Disturbance t-scores/SE. Data was analyzed based on first stage randomization regardless of whether participants were responders or non-responders.
Measure: Mean (Standard Error); unit: T score
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank
Number analyzed (Participants) | 20 | 20
T score
  Baseline | 63.37 (2.5) | 64.160 (2.5)
  Week 4: number analyzed (Participants) | 19 | 19
  Week 4 | 59.46 (2.5) | 59.20 (2.5)
  Week 8: number analyzed (Participants) | 19 | 19
  Week 8 | 56.57 (2.7) | 56.65 (2.6)

6. Secondary Outcome: Cleveland Adolescent Sleepiness Questionnaire (CASQ)
Description: A sixteen-item instrument used to measure daytime sleepiness in adolescents 11-17 years of age.
  Score ranges between 16-80. Higher scores would indicate greater sleepiness
Time Frame: Data Reported on First Stage Randomization of Melatonin vs. Bedtime Bank (Data Collected at: Baseline, Week 4, and Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | First Stage Melatonin | First Stage Bedtime Bank
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 37.70 (7.994) | 41.50 (10.430)
  Week 4: number analyzed (Participants) | 19 | 19
  Week 4 | 35.21 (8.911) | 38.79 (7.052)
  Week 8: number analyzed (Participants) | 19 | 19
  Week 8 | 33.74 (6.723) | 38.42 (8.952)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored by the Data Safety Monitoring Board at the University of Nebraska Medical Center in conjunction with IRB protocols. Adverse event data were collected over the 2 years of the study (2019-2021) from initial consent to end of the trials (approximately 9 weeks).
Description: Adverse events were reported to the DSMB per university protocol. AEs were monitored/assessed according to the intervention received in stage one or stage two. 1 participant had abdominal pain during the baseline week, unrelated to the intervention. 4 participants had mild skin irritation potentially due to wearing the wrist actigraph device (unrelated to intervention). All participants recovered prior to study ending. All-Cause Mortality was not monitored/assessed.
Groups:
- Melatonin Only: Participants in this arm will take 3 mg of melatonin 30 minutes before bedtime.
  Melatonin: Melatonin (liquid, immediate release, 3 mg) 30 minutes before bedtime
- Bedtime Bank Only: Participants in this arm will utilize the Bedtime Bank, a behavioral sleep intervention.
  Bedtime Bank: The Bedtime Bank a novel behavioral sleep intervention, which is based upon contingency contracting and relies on a credit or debt-based system to hold adolescents accountable for maintaining a consistent bedtime and improve total sleep time.
- Combination (Melatonin+Bedtime Bank): Participants in this arm will take 3 mg melatonin 30 minutes before bedtime and utilize the Bedtime Bank, a behavioral sleep intervention.
  Melatonin: Melatonin (liquid, immediate release, 3 mg) 30 minutes before bedtime
  Bedtime Bank: The Bedtime Bank a novel behavioral sleep intervention, which is based upon contingency contracting and relies on a credit or debt-based system to hold adolescents accountable for maintaining a consistent bedtime and improve total sleep time.
Arm/Group | Melatonin Only | Bedtime Bank Only | Combination (Melatonin+Bedtime Bank)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/13
Other Adverse Events (participants affected / at risk) | 3/27 | 2/26 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin Only (N=27) | Bedtime Bank Only (N=26) | Combination (Melatonin+Bedtime Bank) (N=13)
Mild Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 | NA

LIMITATIONS AND CAVEATS:
This K01 study was a pilot feasibility SMART design, which will inform implementation of a future full-scale SMART design to construct adaptive biobehavioral sleep intervention strategies. Pilot SMARTs provide preliminary knowledge about the direction of the effect, and the aims focus on preliminary knowledge; however, conducting formal tests of outcomes or effect size estimation is not justified.

The COVID-19 pandemic began March 2020, and may have impact on study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03730194/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT03730194/ICF_001.pdf